CLINICAL TRIAL: NCT06282237
Title: Clinical Evaluation, Motor Performance and Quality of Life in Patients Affected by Soft Tissue Sarcomas, Undergoing Surgical Treatment: Observational Study
Acronym: 1206
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Sergio Valeri, Principal Investigator, Fondazione Policlinico Universitario Campus Bio-Medico
Other Study IDs: 2022.143
Record Dates: First submitted 2024-01-29; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — Quality of life survey and motor performace survey

SUMMARY:
The main aim of the study is evaluate quality of life and motor performance of patients with soft tissue sarcomas undergoing surgical treatment and post-operative rehabilitation treatment.

Primary objectives:

* Identification of clinical characteristics and motor damage after surgery for soft tissue sarcomas;
* Impact of perioperative treatments and surgery on the quality of life of patients with soft tissue sarcomas;
* Impact of post-operative rehabilitation treatment on quality of life and recovery of motor activity The primary endpoint will be the improvement in the Toronto Extremity Salvage Score (TESS) between T1 (post-surgery) and T3 (at the end of rehabilitation treatment).

Secondary endpoints will be:

1. the evolution over the various timepoints of the selected rating scales (Toronto Extremity Salvage Score, Musculoskeletal Tumor Society Rating Scale, Numerical Rating Scale, Brief Pain Questionnaire, Douleur Neuropathique en 4 Questions, Leeds Assessment of Neuropathic Symptoms and Signs Scale, European Organization for Research and Treatment of Cancer, Quality-of-Life Questionnaire (QLQ)-C30, Short Form Health Survey 36);

• The change in walking performance before and after the rehabilitation treatment.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients affected by primary localized soft tissue sarcoma, candidate to limb/trunk surgery with wide excision or retroperitoneal resection (including resection of the iliopsoas muscle with possible damage to the femoral nerve) with curative intent.

Exclusion Criteria:

* Patients with recurrent tumors;
* patients with metastatic disease;
* patients with palliative surgery;
* patients with amputations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients candidates for surgery for soft tissue sarcoma and undergoing post-operative rehabilitation treatment.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in the Toronto Extremity Salvage Score (TESS) | T0 (1 week before surgery) T1 (1 week post-surgery) and T3 (3 months post-surgery)
  a change in the TESS greater than 7 points

SECONDARY OUTCOMES:
Pain evaluation | T0 (1 week before surgery) T1 (1 week post-surgery) and T3 (3 months post-surgery)
  Brief Pain Questionnaire
Motor performance evaluation | T0 (1 week before surgery) T1 (1 week post-surgery) and T3 (3 months post-surgery)
  Musculoskeletal Tumor Society Rating Scale
Evaluation of Quality of Life | T0 (1 week before surgery) T1 (1 week post-surgery) and T3 (3 months post-surgery)
  Quality-of-Life Questionnaire (QLQ)-C30
Pain evaluation | T0 (1 week before surgery) T1 (1 week post-surgery) and T3 (3 months post-surgery)
  Douleur Neuropathique en 4 Questions
Pain evaluation | T0 (1 week before surgery) T1 (1 week post-surgery) and T3 (3 months post-surgery)
  Leeds Assessment of Neuropathic Symptoms and Signs Scale
Evaluation of Quality of Life | T0 (1 week before surgery) T1 (1 week post-surgery) and T3 (3 months post-surgery)
  Short Form Health Survey 36

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Valeri, Principal Investigator — FPU CampusBioMedico
Locations (1):
- Fondazione Policlinico Campus Biomedico, Roma, Italy

REFERENCES:
- [Result] Bennett M. The LANSS Pain Scale: the Leeds assessment of neuropathic symptoms and signs. Pain. 2001 May;92(1-2):147-57. doi: 10.1016/s0304-3959(00)00482-6. PMID 11323136
- [Result] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Result] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Result] Cacchio A, De Blasis E, Necozione S, Rosa F, Riddle DL, di Orio F, De Blasis D, Santilli V. The Italian version of the lower extremity functional scale was reliable, valid, and responsive. J Clin Epidemiol. 2010 May;63(5):550-7. doi: 10.1016/j.jclinepi.2009.08.001. Epub 2009 Nov 12. PMID 19913388
- [Result] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Result] Davis AM, Wright JG, Williams JI, Bombardier C, Griffin A, Bell RS. Development of a measure of physical function for patients with bone and soft tissue sarcoma. Qual Life Res. 1996 Oct;5(5):508-16. doi: 10.1007/BF00540024. PMID 8973131
- [Result] den Hollander D, Van der Graaf WTA, Fiore M, Kasper B, Singer S, Desar IME, Husson O. Unravelling the heterogeneity of soft tissue and bone sarcoma patients' health-related quality of life: a systematic literature review with focus on tumour location. ESMO Open. 2020 Oct;5(5):e000914. doi: 10.1136/esmoopen-2020-000914. PMID 33082266
- [Result] Gerrand C, Furtado S. Issues of Survivorship and Rehabilitation in Soft Tissue Sarcoma. Clin Oncol (R Coll Radiol). 2017 Aug;29(8):538-545. doi: 10.1016/j.clon.2017.04.001. Epub 2017 Apr 22. PMID 28442210
- [Result] Kask G, Repo JP, Tukiainen EJ, Blomqvist C, Barner-Rasmussen I. Soft Tissue Sarcoma of Lower Extremity: Functional Outcome and Quality of Life. Ann Surg Oncol. 2021 Oct;28(11):6892-6905. doi: 10.1245/s10434-021-09774-6. Epub 2021 Mar 19. PMID 33740199
- [Result] Kask G, Barner-Rasmussen I, Repo JP, Kjaldman M, Kilk K, Blomqvist C, Tukiainen EJ. Functional Outcome Measurement in Patients with Lower-Extremity Soft Tissue Sarcoma: A Systematic Literature Review. Ann Surg Oncol. 2019 Dec;26(13):4707-4722. doi: 10.1245/s10434-019-07698-w. Epub 2019 Aug 12. PMID 31407171
- [Result] Ogura K, Uehara K, Akiyama T, Shinoda Y, Iwata S, Tsukushi S, Kobayashi E, Hirose T, Yonemoto T, Endo M, Tanzawa Y, Nakatani F, Kawano H, Tanaka S, Kawai A. Minimal clinically important differences in Toronto Extremity Salvage Score for patients with lower extremity sarcoma. J Orthop Sci. 2020 Mar;25(2):315-318. doi: 10.1016/j.jos.2019.03.022. Epub 2019 Apr 16. PMID 31000377
- [Result] Padua L, Briani C, Jann S, Nobile-Orazio E, Pazzaglia C, Morini A, Mondelli M, Ciaramitaro P, Cavaletti G, Cocito D, Fazio R, Santoro L, Galeotti F, Carpo M, Plasmati R, Benedetti L, Schenone A, Marchettini P, Cruccu G. Validation of the Italian version of the Neuropathic Pain Symptom Inventory in peripheral nervous system diseases. Neurol Sci. 2009 Apr;30(2):99-106. doi: 10.1007/s10072-009-0025-y. Epub 2009 Feb 6. PMID 19198756
- [Result] Sartorio F, Moroso M, Vercelli S, Bravini E, Medina ME, Spalek R, Ferriero G. [CROSS-CULTURAL ADAPTATION, AND VALIDITY OF THE ITALIAN VERSION OF THE UPPER LiMB FUNCTIONAL INDEx (ULFI-I)]. G Ital Med Lav Ergon. 2015 Apr-Jun;37(2):115-9. Italian. PMID 26364445
- [Result] Rossi L, Boffano M, Comandone A, Ferro A, Grignani G, Linari A, Pellegrino P, Piana R, Ratto N, Davis AM. Validation process of Toronto Exremity Salvage Score in Italian: A quality of life measure for patients with extremity bone and soft tissue tumors. J Surg Oncol. 2020 Mar;121(4):630-637. doi: 10.1002/jso.25849. Epub 2020 Jan 19. PMID 31957034
- [Result] Van Seventer R, Vos C, Meerding W, Mear I, Le Gal M, Bouhassira D, Huygen FJ. Linguistic validation of the DN4 for use in international studies. Eur J Pain. 2010 Jan;14(1):58-63. doi: 10.1016/j.ejpain.2009.01.005. Epub 2009 Mar 17. PMID 19282208
- [Result] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Derived] Demofonti A, Brunetti B, Germanotta M, Coppola MM, Falchini F, Valeri A, Tenna S, Valeri S, Aprile IG. Effects of a tailored rehabilitation treatment in lower limb Soft Tissue Sarcomas reconstruction: a case series. J Neuroeng Rehabil. 2026 Jan 21. doi: 10.1186/s12984-026-01878-y. Online ahead of print. PMID 41566361